CLINICAL TRIAL: NCT06698237
Title: The Effects of Delayed Versus Immediate Cold-water Immersion on Exercise Performance Recovery and Postprandial Plasma Aminoacidemia Following Exercise and Protein Consumption in Athletes
Brief Title: The Effects of Cold-water Immersion on Exercise Performance Recovery and Postprandial Plasma Aminoacidemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Associate Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-01-046
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-04

CONDITIONS: Sport Recovery; Aminoacidemia; Cold-water Immersion
Keywords: Cold-water immersion; Protein; Performance; Athlete; Exercise physiology; Nutrition; Exercise; Resistance training; Sport recovery; Aminoacidemia; cold-therapy; strength training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized crossover design, 12 participants (6 male and 6 female)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CWI_0 (Experimental): immediate cold-water immersion
  Interventions: Other: immediate cold-water immersion
- CWI_3 (Experimental): 3 hour delayed cold water immersion
  Interventions: Other: delayed cold-water immersion
- THERM (Active Comparator): immediate thermoneutral water immersion
  Interventions: Other: immediate thermoneutral water immersion

INTERVENTIONS:
Other: immediate cold-water immersion — immediate 10 minute water immersion in 10 degree Celsius
  Arms: CWI_0
Other: delayed cold-water immersion — 3 hour delayed 10 minute water immersion in 10 degree Celsius
  Arms: CWI_3
Other: immediate thermoneutral water immersion — immediate 10 minute water immersion in 35 degree Celsius
  Arms: THERM

SUMMARY:
In order to optimize sports performance, high-level athletes are required to manage conflicting training objectives, which often result in periods of high-volume training. These athletes need to perform heavy resistance training sessions to promote physiological adaptations, which consequently induce fatigue. Yet, they need to minimize fatigue to perform subsequent high-quality training sessions often within the same day. To support these training endeavours, a high-quality dietary regimen and adequate protein consumption is deemed to be an essential component of an athlete's recovery plan, as it has been shown to support muscle recovery and reduce muscle inflammation following exercise. Indeed, current sports nutrition recommendations advocate for the consumption of dietary protein and carbohydrate after exercise to promote tissue repair and replenish muscle energy stores (glycogen). Additionally, previous research has shown how water immersion therapies post-exercise may alleviate fatigue and restore performance. However, little is known about how different temperatures, as well as timing of cold-water immersion can support performance recovery in a population of athletes adhering to contemporary post-exercise nutrition recommendations. The objective of this project is to investigate the effects of timing of cold-water immersion relative to exercise on performance recovery within the same day, as well as to investigate whether cold water immersion augments blood amino acid concentrations after exercise and protein intake.

DETAILED DESCRIPTION:
In the 48-hours prior to testing visits, participants will need to fill out a dietary log 2 days before the first visit and replicate their diet before the second and third visit. Participants will also be asked to adhere to the same exercise routine in order to replicate exercise behaviours for all testing days. Testing sessions will be separated by a minimum of seven days but not more than 30 days. The female participants with a regular menstrual cycle will only be tested during the follicular phase (from day one of menstruation and lasts fourteen days) to ensure a standardized hormone level. Each testing day will begin in the morning. Participants will arrive in the laboratory in an overnight fasted state and begin by ingesting a telematic pill and then consume a standardized carbohydrate rich breakfast drink. Afterwards, the athlete will complete the performance tests, which will include five counter-movement jumps, five drop jump, five squat jumps, one 5-second maximal voluntary isometric contraction (MVIC) of the knee-extensors, eight 1-second maximal voluntary isometric contractions (MVIC) of the knee extensors, five maximal isokinetic contractions at three different angular velocities (60, 180, and 240°/s). Then, they will perform the resistance training protocol, consisting of ten sets on the leg press at 65% 1RM. The 1st and 10th sets will be taken to failure. Sets 2 to 9 will be performed at 10 repetitions each. Between set 1 and set 2, they will perform 30 depth drops. The rest time between sets will be two minutes. Immediately post-training, participants will be asked to repeat the same performance tests. They will then be provided with a protein and carbohydrate drink (25 g of whey protein and 45 g of carbohydrate) that will be consumed within 5 minutes. During the experimental visit, 11 blood samples will be collected relative to the water immersion (T = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, and 300 min), and subsequently analysed for postprandial plasma amino acid concentration. The consumption of the beverage will be followed by an 10-minute mid-clavicular immersion in either CWI (10°C) that is immediate (CWI_0), delayed for 3-hours (CWI_3), or an immediate thermoneutral bath (35°C) (THERM). Following the final blood draw (T = 300 min), the performance tests will be performed one last time to evaluate recovery from the strength training. The participant will be asked to fill out the Short Recovery and Stress Scale (SRSS) that measures recovery and stress across emotional, mental, physical, and overall dimensions using eight items before each testing session. They will also be asked to fill out a visual analogue scale (VAS) regarding subjective appetite sensations at the same time as every blood sample. Furthermore, skin and core body temperatures will be monitored throughout the experiment. At the end of each of the experimental visits, the participants will receive an ad libitum pasta meal to measure energy intake. The participants will be instructed to eat until they are comfortably full within 30 minutes. The amount of food consumed will be recorded to calculate the energy intake of each participant. Participants will also need to complete a questionnaire the 24 and 48 hours after each testing session to assess their level of delayed onset muscle soreness. Following the final testing session, participants will be invited to complete a belief questionnaire, aimed at gauging their perceived effectiveness of the recovery conditions they were subjected to.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this study, a participant must meet all the following criteria:

1. Healthy adult between 18 - 40 years (inclusive).
2. Individual with a BMI between >18.5 and <30 kg/m2 (inclusive).
3. Individual who is in good general health (no uncontrolled diseases or conditions).
4. individual with a history of regular resistance training ≥2 per week for the past six-months.
5. Individual who is currently competing at the varsity, provincial, national or international level in their respective sport.
6. Individual who is free from any musculoskeletal injuries and/or conditions that might affect their ability to perform resistance exercises or undergo cold-water immersion.
7. Individual who has maintained stable use of medication and/or supplements, stable dietary and lifestyle habits, and stable body weight (weight loss or gain <3 kg), for the last three-months prior to screening.
8. Individual who agrees to maintain usual training habits between sessions.

Exclusion Criteria

1. Individual who is lactating, pregnant or planning to become pregnant during the study.
2. Females with irregular menstrual cycles (defined as outside 24-38 days cycle range, based on self-reports).
3. Individual who adheres to a diet (e.g., vegan diet) that restricts consumption of dairy products.
4. Has a known sensitivity, intolerability, or allergy to any of the study products or their excipients (i.e., lactose intolerant).
5. Weight loss or gain > 3 kg in the 3 months prior to study visit 1.
6. Currently or planning to be on a weight loss regimen during the study.
7. Recent (within 2 weeks of screening visit) history of an episode of acute GI illness such as nausea/vomiting or diarrhea.
8. Have a history of irritable bowel disease (IBS), inflammatory bowel disease (IBD, including ulcerative colitis and Crohn's disease), functional constipation or diarrhea (defined by the Rome IV diagnostic criteria), celiac disease, malabsorption, gastroparesis, diverticulosis, gastric or duodenal ulcers, pancreatitis, or eating disorder; or have a history of intestinal surgery (excluding appendectomy or herniorrhaphy) or bariatric surgery.
9. Have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and/or digestion (e.g., history of bowel obstruction).
10. Participated in upper gastrointestinal endoscopy and/or colonoscopy or preparation within 3 months prior to screening visit.
11. Diagnosed with hypercholesterolemia or hypertriglyceridemia (i.e., elevated fasting low- density lipoprotein (LDL) (≥ 135 mg·dL-1; ≥ 3.5 mmol·L-1) or elevated triglycerides (≥ 150 mg·dL-1; ≥1.7 mmol·L-1).
12. Has a history of heart disease/cardiovascular disease, uncontrolled hypertension (≥ 140 systolic or ≥ 90 diastolic mmHg), kidney disease (dialysis or renal failure), hepatic impairment or disease.
13. Is Type I or Type II diabetic or pre-diabetic [i.e., elevated fasting blood glucose levels (≥ 100 mg·dL-1; ≥ 5.6 mmol·L-1) and/or elevated hemoglobin A1c (≥ 6.0%)].
14. Has a history of liver or gallbladder disease or stomach ulcers.
15. Has a positive medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorders and/or immunocompromised (e.g., HIV/AIDS).
16. Diagnosed with cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to the screening visit, or any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential participant at risk because of participation in the study, or influences the results or the potential participant's ability to participate in the study.
17. Major surgery in 3 months prior to screening or planned major surgery during the study.
18. History of alcohol or substance abuse (including cannabinoids) in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program).
19. Current or previous tobacco use within the last 6 months.
20. Self-report of blood donation totaling between 101 mL to 449 mL of blood within 30 days prior to screening or a blood donation of more than 450 mL within 56 days prior to baseline.
21. Self-report of donating plasma (e.g., plasmapheresis) within 14 days prior to screening.
22. Any other active or unstable medical conditions or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — cis-male and cis-female
Enrollment: 12 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prolonged maximum voluntary isometric contraction of the knee extensors peak force | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform one five-second maximum voluntary isometric contraction of the knee extensors on an isometric dynamometer at a 60° angle of the knee joint. The force-time profile will be used to derive the peak force (Newton)

SECONDARY OUTCOMES:
postprandial plasma total amino acid concentration incremental area-under-the-curve | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma branched chain amino acid concentration incremental area-under-the-curve | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma essential amino acid concentration incremental area-under-the-curve | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma leucine concentration incremental area-under-the-curve | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  leucine at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
Postprandial plasma glucose concentration incremental area-under-the-curve | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Plasma glucose at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) (mmol/L·300 minutes).
Postprandial plasma insulin concentration incremental area-under-the-curve | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minute in the post-prandial period
  Plasma insulin at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minute) (pmol/L·300 minute).
postprandial plasma total amino acid time to concentration maximum | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma branched chain amino acid time to concentration maximum | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma essential amino acid time to concentration maximum | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma leucine time to concentration maximum | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  leucine at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) (umol/L)
postprandial plasma total amino acid concentration maximum | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma branched chain amino acid concentration maximum | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma essential amino acid concentration maximum | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma leucine concentration maximum | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  leucine at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) (umol/L)
postprandial plasma total amino acid time tracking response | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma branched chain amino acid time tracking response | 120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma essential amino acid time tracking response | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined) at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) umol/L
postprandial plasma leucine time tracking response | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  leucine at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) (umol/L)
Postprandial plasma glucose time tracking response | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Plasma glucose at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) (mmol/L·300 minutes).
Postprandial plasma insulin time tracking response | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Plasma insulin at 11 timepoints (t = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes) (pmol/L·300 minutes).
Postprandial appetite sensation scores time tracking response | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Participants will be asked to complete visual analog scales (VAS) for measurements of appetite sensations at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes). Five sensations related to appetite are queried by VAS (i.e., "How hungry are you?", "How full are you?", "How satiated are you?", "How strong is your desire to eat?" on a scale from "Not at all" to "Extremely"; and "How much do you think you could (or would want to) eat right now" on a scale from "nothing at all" to "a very large amount"). Outcomes are measured in millimeters (mm) along a 100-mm horizontal line
Postprandial appetite sensation incremental-area-under-the-curve | -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes in the post-prandial period
  Participants will be asked to complete visual analog scales (VAS) for measurements of appetite sensations at 11 timepoints (time = -120, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes). Five sensations related to appetite are queried by VAS (i.e., "How hungry are you?", "How full are you?", "How satiated are you?", "How strong is your desire to eat?" on a scale from "Not at all" to "Extremely"; and "How much do you think you could (or would want to) eat right now" on a scale from "nothing at all" to "a very large amount"). Responses are measured in mm·300 minutes.
Ad libitum food energy intake | assessed 300 minutes after protein intake
  The ad libitum test meal will contain 562 kJ per 100 g with 20% energy from protein, 65% energy from carbohydrate, and 15% energy from fat. The participants will be provided with approximately 1 kg of the test meal on a plate with utensils. Participants will be instructed to "eat as much or as little as desired until feeling "comfortably full" within 30 minutes. The meal will be weighed before consumption and remaining contents will be weighed after achieving comfortable fullness to calculate the energy intake. The outcome will be measure in kilojoules (kJ).
Countermovement jump | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five countermovement jumps on a force plate. The jump height derived from impulse (centimeter), maximum force developed (Newton), maximum rate of force development (Newton/second) will be collected for each of the five jumps. The change from baseline will be reported.
Intermitted Maximum voluntary isometric contraction of the knee extensors peak force | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform eight one-second maximum voluntary isometric contraction of the knee extensors on an isometric dynamometer at a 60° angle of the knee joint. The force-time profile will be used to derive the peak force (Newton)
Maximal Leg Press Strength | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform repetitions till failure using a weight equivalent to 65% of their maximum strength. The total number of repetitions completed, the average velocity, peak velocity and work of the repetitions will be recorded and the change from baseline in these values will be reported.
recovery-stress state | 2 hours prior to protein intake, immediately prior to protein intake, 5 hours post protein intake, 24 hours and 48 hours post training
  The participant will be asked to fill out the Short Recovery and Stress Scale (SRSS) that measures recovery and stress across emotional, mental, physical, and overall dimensions using eight items.
Delayed onset muscle soreness | reported 120 minutes prior to water immersion, 300 minutes post protein intake, and at 24 hours and 48 hours post testing.
  Participants will be asked to complete visual analog scales (VAS) for a measurement of muscle soreness on a scale from "normal" to "extremely sore"). Outcome is measured in millimeters (mm) along a 100-mm horizontal line. Data will be reported 120 minutes prior to water immersion, 300 minutes post protein intake, and at 24 hours and 48 hours post testing.
Serum concentrations of systemic cytokines | -120, 0, 30, 60, 120, 180, 240, 300 minutes in the post-prandial period
  time-course concentration of serum concentrations of systemic cytokines IL-6, IL-8, IL-1B, TNF-α, IL-10 (pg/ml) at 8 timepoints (time = -120, 0, 30, 60, 120, 180, 240, 300 minutes).
Time-course of heart rate | Data will be reported during the resistance -90 to -30 minutes and during water immersion 0 minutes to 10 minutes or 180 minutes to 190 minutes
  The participants heart rate will be monitored using a heart rate monitor. The average heart rate during resistance training and during water immersion will be reported.
Time-course of skin temperature | 0 to 5 hours post water immersion.
  The participants skin temperature will be monitored using sensors that can record temperature data over time) (sampling frequency = 30 seconds). The sensors will be placed on the sternum, forearm, thigh and calf. The outcome is measured in degrees Celsius. Data will be reported every 15 minutes following water immersion and every hour before and after following water immersion.
Core temperature | 0 to 5 hours post water immersion
  The participants core temperature will be monitored using telemetric thermometer pill that will be ingested upon arrival at the laboratory (sampling frequency = 30 seconds). The outcome is measured in degrees Celsius. Data will be reported every 5 minutes during water immersion, every 15 minutes for 1 hour following water immersion. Data will otherwise be reported every hour.
Incidence of adverse events | 0-6 hours post water immersion
  Number of participants with adverse events
Prolonged maximum voluntary isometric contraction of the knee extensors total work | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake
  The participant will be asked to perform one five-second maximum voluntary isometric contraction of the knee extensors on an isometric dynamometer at a 60° angle of the knee joint. The force-time profile will be used to derive the area under the curve (N·5 s). The change from baseline will be reported.
Prolonged maximum voluntary isometric contraction of the knee extensors rate of force developpment | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake
  The participant will be asked to perform one five-second maximum voluntary isometric contraction of the knee extensors on an isometric dynamometer at a 60° angle of the knee joint. The force-time profile will be used to derive the rate of force development (N/s). The change from baseline will be reported.
Intermitted Maximum voluntary isometric contraction of the knee extensorsIntermitted Maximum voluntary isometric contraction of the knee extensors rate of force development | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake
  The participant will be asked to perform eight one-second maximum voluntary isometric contraction of the knee extensors on an isometric dynamometer at a 60° angle of the knee joint. The force-time profile will be used to derive the rate of force development (N/s) for each of the eight contractions. The change from baseline will be reported.
Isokinetic testing of the knee extensors 60°/second peak torque | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 60°/second. The force-time profile will be used to derive the peak torque (Newton-metre) change from baseline will be reported.
Isokinetic testing of the knee extensors 180°/second peak torque | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 180°/second. The force-time profile will be used to derive the peak torque (Newton-metre) change from baseline will be reported.
Isokinetic testing of the knee extensors 240°/second peak torque | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 240°/second. The force-time profile will be used to derive the peak torque (Newton-metre) change from baseline will be reported.
Isokinetic testing of the knee extensors 60°/second total work | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 60°/second. The force-time profile will be used to derive the total work (Joules). The change from baseline will be reported.
Isokinetic testing of the knee extensors 180°/second total work | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 180°/second. The force-time profile will be used to derive the total work (Joules). The change from baseline will be reported.
Isokinetic testing of the knee extensors 240°/second total work | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 240°/second. The force-time profile will be used to derive the total work (Joules). The change from baseline will be reported.
Isokinetic testing of the knee extensors 60°/second average power | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 60°/second. The force-time profile will be used to derive the average power (Watts) The change from baseline will be reported.
Isokinetic testing of the knee extensors 180°/second average power | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 180°/second. The force-time profile will be used to derive the average power (Watts) The change from baseline will be reported.
Isokinetic testing of the knee extensors 240°/second average power | 120 minutes prior to water immersion, immediately prior to water immersion, 300 minutes post protein intake.
  The participant will be asked to perform five isokinetic contractions of the knee extensors at 240°/second. The force-time profile will be used to derive the average power (Watts) The change from baseline will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No